CLINICAL TRIAL: NCT02201225
Title: A Methodology Study to Evaluate a Sitting Knee Measuring Device in Assessing Growth in Indian Children Aged 6 to 12 Years Receiving Nutritional Supplement With or Without Micronutrient Fortification
Brief Title: A Methodology Study to Evaluate a Sitting Knee Measuring Device in Assessing Growth in Indian Children.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201133; RH01817 (Other: GSK)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Nutritional Status
MeSH Terms: interventions — Dietary Supplements; Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplement with micronutrient (Active Comparator): Nutritional supplement powder with micronutrients packed as 27 g individual sachet, administered orally as a single serve twice daily
  Interventions: Dietary Supplement: Nutritional supplement with micronutrient
- Nutritional supplement without micronutrient (Sham Comparator): Nutritional supplement powder without micronutrients packed as 27 g individual sachet, administered orally as a single serve twice daily
  Interventions: Dietary Supplement: Nutritional supplement without micronutrient

INTERVENTIONS:
Dietary Supplement: Nutritional supplement with micronutrient — Nutritional supplement powder with micronutrients packed as 27 g individual sachet, administered orally as a single serve
  Arms: Nutritional supplement with micronutrient
Dietary Supplement: Nutritional supplement without micronutrient — Nutritional supplement powder without micronutrients packed as 27 g individual sachet, administered orally as a single serve
  Arms: Nutritional supplement without micronutrient

SUMMARY:
This methodology study will evaluate the sensitivity in using sitting knee digital caliper to measure changes in sitting knee length from over a 12-week study period amidst children in the age of 6 to 12 years in a community-based study in children ages 6 to 12 years who are receiving nutritional supplementation with micronutrients or without micronutrients.

ELIGIBILITY:
Inclusion Criteria:

* Children (participants), both boys and girls, aged 6 to 12 years.
* Participant height to be within the 25th to the 75th percentile of the standard height average in Indian children population
* Participant will agree not to take any other nutritional supplements products during the study except the trial supplement

Exclusion Criteria:

* Participant has any of the following medical conditions: Genetic disorders, chronic disease, metabolic disorders, endocrine disorders, immobilisation, and miscellaneous
* Participant who in the past 6 months has used dietary or nutritional supplements with micronutrient fortification, or any form of dietary or herbal supplement intended to increase micronutrient intake, at a frequency of greater than 3-4times per month.
* Participant receiving any supplements (such as calcium, iron and/or multivitamin at the time of screening).
* Children (Participant) in Care are not allowed to participate in the study.
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Health conditions that would affect food metabolism including the following food allergies, kidney disease, liver disease, and/or gastrointestinal diseases (e.g. irritable bowel syndrome, celiac disease, peptic ulcers).
* Use of concomitant medications that, in the opinion of the Principal Investigator (PI), might interfere with the outcome of the study or increases the risk of the participant, including corticosteroids (systemic or inhaled) and any medication for any behaviour-related disorders and/or stimulants.
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder, including history of alcohol or substance abuse, that would make the participant unlikely to fully complete the study or any condition that presents undue risk from the study product or procedures in the opinion of the PI/medical examiner.
* Clinical Study/Experimental Medication: Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Personnel: Currently, the participant's parents/legal guardian is an employee of the Sponsor or the study or members of their immediate family.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in bone growth, as measured by sitting knee length caliper. | Baseline to Week 12
  To evaluate the sensitivity of a sitting knee digital caliper to measure changes in sitting knee length from Baseline to Week 12 in a community-based study in the presence of nutritional supplementation with or without micronutrients.

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in Z-score based on the standing height | Baseline-Week 12
  Comparison of standing height and sitting knee height to asses growth
Change from Baseline to Week 8 in bone growth, as measured by sitting knee length digital caliper | Baseline-Week 8
  To assess the relationship between changes from Baseline to Week 8 in sitting knee length and standing height in the presence of nutritional supplementation with or without micronutrients

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangalore, India

REFERENCES:
- See also: Results for Study 201133 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/201133?search=study&study_ids=201133#rs